CLINICAL TRIAL: NCT02317627
Title: A Phase 2, Open-Label, Dose-finding Study to Evaluate the Safety, Tolerability, and Activity of KD025 in Subjects With Psoriasis Vulgaris Who Failed First-line Therapy
Brief Title: Phase 2, Open-label, Study of KD025 in Subjects With Psoriasis Vulgaris Who Failed First-line Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kadmon Corporation, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KD025-206
Record Dates: First submitted 2014-12-10; First posted 2014-12-16 (Estimated); Results first posted 2021-11-01 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — KD025; belumosudil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): KD025 400 mg QD PO for 12 weeks
  Interventions: Drug: KD025
- Cohort 2 (Experimental): KD025 200 mg BID PO for 12 weeks
  Interventions: Drug: KD025
- Cohort 3 (Experimental): KD025 400 mg BID PO for 12 weeks
  Interventions: Drug: KD025

INTERVENTIONS:
Drug: KD025
  Other Names: SLx-2119; belumosudil

SUMMARY:
This study was performed to evaluate the safety, tolerability, activity, pharmacokinetics (PK), and daily dose regimen of KD025 administered orally (PO) for 12 weeks to subjects with psoriasis vulgaris who failed at least one line of systemic therapy.

DETAILED DESCRIPTION:
Study KD025-206 was a phase 2, open-label, dose-finding, safety, tolerability, activity, and PK study of KD025 in subjects with psoriasis who had failed at least 1 line of systemic therapy or phototherapy.

Subjects received KD025 PO for 12 weeks. Planned enrollment was 36 subjects in 3 cohorts, 12 subjects per cohort:

* Cohort 1 (12 subjects): KD025 400 mg once daily (QD) PO for 12 weeks
* Cohort 2 (12 subjects): KD025 200 mg PO twice daily (BID) for 12 weeks
* Cohort 3 (12 subjects): KD025 400 mg BID PO for 12 weeks

Subjects were initially enrolled simultaneously in Cohort 1 and Cohort 2 according to a randomization schedule, with safety reviewed before any subjects. If safety guidelines were met, Cohort 3 was added to explore the efficacy and safety of KD025 at a dose of 400 mg PO BID.

Subjects underwent safety evaluations: medical history evaluations; physical examinations (PEs); vital sign measurements; weight measurements; adverse event (AE) assessments; concomitant medication assessments; blood sample collection for hematology, chemistry, and coagulation; lipid panel; thyroid-stimulating hormone; measurements of antinuclear antibody; anti-double-stranded deoxyribonucleic acid; Complement C; antiphospholipid antibody; liver ultrasound (US); pregnancy testing for females of childbearing potential; PK sampling (subset of subjects only); urinalysis; and electrocardiogram (ECG).

Subjects underwent efficacy evaluations: Psoriasis Area and Severity Index (PASI) scoring; Physicians Global Assessment (PGA) scoring; and Dermatologic Life Quality Index (DLQI) scoring.

Subjects participating in PK sampling were admitted to the clinic on Month 1 Day 1 (M1D1) for PK procedures and were discharged on M2D2. Blood samples for PK analyses were collected on M2D1 and Month 3 Day 1 (M3D1) on an outpatient basis. Subjects were not to take their morning dose until after blood samples were drawn.

A Follow-Up visit occurred 30 ± 3 days after the last dose of study drug.

The endpoints for efficacy were PASI, PGA, and DSQI scores.

1. Psoriasis Area and Severity Index (PASI): The PASI is a measure of the psoriasis disease severity using the average redness, thickness, and scaliness of the lesions (each graded on a 0 to 4 scale), which is weighted by the area of involvement. The PASI combines the assessment of the severity of lesions and the area affected into a single score ranging from 0 (no disease) to 72 (maximal disease).
2. Physicians Global Assessment (PGA): The relative PGA documents the physician's assessment of the subject's psoriasis status. Consideration was given to the percent of body involvement as well as overall induration, scaling, and erythema. The PGA was assessed relative to baseline condition and defined as: (1) clear; (2) excellent; (3) good; (4) fair; (5) poor; and (6) worse.
3. Dermatology Life Quality Index (DLQI): The DLQI is a skin disease-specific instrument designed to assess the impact of the disease on a subject's quality of life (QOL). It is a 10-item questionnaire that assesses 6 different aspects of quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. Possible DLQI scores range from 0 (no detectable impairment on a subject's QOL) to 30 (extremely large effect on a subject's QOL).

Safety was assessed by standard clinical and laboratory tests (hematology, serum chemistry, and urinalysis), PEs, and reporting of treatment-emergent adverse events (TEAEs). Toxicity grades were defined using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. In addition, subjects had liver ultrasound and liver functioning testing assessed for possible steatosis.

Blood samples for determination of PK plasma concentrations of KD025 and its metabolites were collected for maximum concentration (Cmax); time of maximum concentration (Tmax); area under the concentration-time curve (AUC) at 0 to 24 hours, 0 to last, and 0 to infinity (0 to 24, 0 to last, 0 to infinity [inf]); half-life (t1/2); and accumulation ratio (metabolic-to-parent drug ratio).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent prior to the performance of any study specific procedures
* Diagnosis of moderately severe plaque psoriasis that has been moderately stable for 6 months and failed at least 1 line of systemic or phototherapy and is a candidate for additional systemic therapy
* PASI of ≥ 12 within the 24-hour period prior to the first dose of study drug
* At least 10% of body surface area affected by plaque psoriasis within the 24-hour period prior to the first dose of study drug
* Willing to avoid tanning devices
* Willing to forgo other systemic and topical treatments for psoriasis during the course of the study
* Adequate bone marrow function: absolute neutrophil count > 1500/mm^3; hemoglobin > 9.0 g/dL; platelets > 100,000/mm^3
* Negative urine pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug
* Agree to use a highly effective method of birth control (< 1% per year failure rate) during the study and for 1 month after the termination of the study. Effective birth control included implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence, or vasectomized partner
* Willing to complete all study measurements and assessments in compliance with the protocol

Exclusion Criteria:

* Non-plaque or drug-induced (antimalarials, lithium) psoriasis (If subject is taking angiotensin II receptor blockers or beta blockers doses had to be stable for 6 months prior to study entry)
* Use of corticosteroid or immunosuppressive therapy within 4 weeks prior to study entry except for Class 5 or weaker topical corticosteroids or immunosuppressive therapies to the face, groin, or scalp.
* Use of methotrexate, acitretin, or cyclosporine within 4 weeks prior to study entry
* Use of phototherapy within 4 weeks prior to study entry
* Use of biologic therapies, including antibodies to IL-17, within 3 months prior to study entry
* Concomitant condition requiring treatment with moderate to high dose steroids in the 12 weeks prior to screening
* Viral, fungal, or bacterial skin infection
* Pregnant or lactating
* History of gastrointestinal (GI) surgery including bariatric surgery, or any GI condition that might interfere with drug absorption
* Currently participating in another study with an investigational drug or within 28 days of study entry
* History or other evidence of severe illness or any other conditions that would make the subject, in the opinion of the investigator, unsuitable for the study (such as poorly controlled psychiatric disease or coronary artery disease)
* Regular and excessive use of alcohol within the 2 years prior to study entry defined as alcohol intake > 14 drinks per week in a man or > 7 drinks per week in a woman. Approximately 10 g of alcohol equals one "drink" unit. One unit equals 1 ounce of distilled spirits, one 12-ounce beer, or one 4-ounce glass of wine
* History or presence of any of the following:

  1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.0 × the upper limit of normal (ULN) at screening. (Subjects with an isolated AST elevation of any magnitude, or a ratio of AST:ALT > 1.5 interviewed regarding use of alcohol, have levels repeated and participation in the study should be discussed with the medical monitor.)
  2. Renal disease and/or serum creatinine > 1.5 × ULN at screening
* QTc(F) interval (QT interval data corrected using Fridericia's formula) > 450 msec at the screening or predose ECG
* Previous exposure to KD025 or known allergy/sensitivity to KD025 or any other ROCK-2 inhibitor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Arrowhead Health Centers, Glendale, Arizona
  - Southern California Dermatology, Inc., Santa Ana, California
  - Shondra L. Smith, Lake Charles, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Clinical Studies Group, LLC, Henderson, Nevada
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - High Point Clinical Trials Center, High Point, North Carolina
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Metroplex Clinical Research Center (MCRC), Dallas, Texas

REFERENCES:
- [Background] Zanin-Zhorov A, Weiss JM, Trzeciak A, Chen W, Zhang J, Nyuydzefe MS, Arencibia C, Polimera S, Schueller O, Fuentes-Duculan J, Bonifacio KM, Kunjravia N, Cueto I, Soung J, Fleischmann RM, Kivitz A, Lebwohl M, Nunez M, Woodson J, Smith SL, West RF, Berger M, Krueger JG, Ryan JL, Waksal SD. Cutting Edge: Selective Oral ROCK2 Inhibitor Reduces Clinical Scores in Patients with Psoriasis Vulgaris and Normalizes Skin Pathology via Concurrent Regulation of IL-17 and IL-10. J Immunol. 2017 May 15;198(10):3809-3814. doi: 10.4049/jimmunol.1602142. Epub 2017 Apr 7. PMID 28389592

RESULTS

PARTICIPANT FLOW:
Groups:
- 400 mg QD: Belumosudil 400 mg administered orally (PO) once daily (QD) for 12 weeks
- 200 mg BID: Belumosudil 200 mg administered PO twice daily (BID) for 12 weeks
- 400 mg BID: Belumosudil 400 mg administered PO BID for 12 weeks
Period: Overall Study
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID
Started | 13 | 13 | 12
Completed | 11 | 8 | 8
Not Completed | 2 | 5 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Stopped by Investigator | 0 | 1 | 0
Not completed — Adverse Event | 0 | 2 | 3
Not completed — Non-compliance with study drug | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) defined as all subjects enrolled in the study
Groups:
- 400 mg QD: Belumosudil 400 mg PO QD for 12 weeks
- 200 mg BID: Belumosudil 200 mg PO BID for 12 weeks
- 400 mg BID: Belumosudil 400 mg PO BID for 12 weeks
- Total: Total of all reporting groups
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Total
Number analyzed (Participants) | 13 | 13 | 12 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (10.32) | 46.5 (11.92) | 50.5 (10.26) | 47.1 (10.86)
Age, Continuous [Median (Full Range); unit: years] | 46.0 [29 to 60] | 45.0 [25 to 67] | 54.5 [30 to 64] | 47.5 [25 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 4 | 15
  Male | 8 | 7 | 8 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 6 | 15
  Not Hispanic or Latino | 8 | 9 | 6 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 11 | 12 | 12 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
BMI (body mass index)--Mean [Mean (Standard Deviation); unit: kg/m^2] | 34.42 (7.132) | 32.81 (7.747) | 32.65 (10.582) | 33.31 (8.362)
BMI--Median [Median (Full Range); unit: kg/m^2] | 35.70 [22.2 to 45.4] | 31.40 [23.4 to 51.4] | 30.35 [22.7 to 63.8] | 31.50 [22.2 to 63.8]
Psoriasis Area and Severity Index (PASI) Score--Mean [Mean (Standard Deviation); unit: Units on a scale] — The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign is assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.
  Units on a scale | 21.0 (10.85) | 18.3 (8.51) | 20.3 (7.24) | 19.8 (8.87)
PASI--Median [Median (Full Range); unit: Units on a scale] — The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign is assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.
  Units on a scale | 18.0 [12.8 to 52.8] | 16.2 [12.0 to 42.0] | 18.5 [12.9 to 32.2] | 17.3 [12.0 to 52.8]
Physician Global Assessment (PGA) [Count of Participants; unit: Participants] — The Physician Global Assessment (PGA) documents the physician's assessment of the subject's psoriasis and is assessed relative to baseline conditions. The PGA rating is from 1-6, where 1 = 100% clearing of psoriasis (clear), 5 = 0 to 24% clearing (little or no change), and 6 = worse.
  Participants
    Clear (100%) | 0 | 0 | 0 | 0
    Excellent (75% to 99%) | 0 | 0 | 0 | 0
    Good (50% to 74%) | 0 | 0 | 0 | 0
    Fair (25% to 49%) | 1 | 5 | 2 | 8
    Poor (0% to 24%) | 12 | 6 | 7 | 25
    Worse | 0 | 2 | 3 | 5
Dermatology Quality Life Index (DQLI)--Mean [Mean (Standard Deviation); unit: Units on a scale] — The Dermatology Life Quality Index (DLQI) is a skin disease-specific instrument designed to assess the impact of the disease on a subject's quality of life. The scale range is 0 to 30: 0-1=no effect on subject's life; 2-5=small effect; 6-10= moderate effect; 11-20=very large effect; 21-30=extremely large effect.
  Units on a scale | 14.6 (6.79) | 14.2 (6.39) | 10.3 (7.77) | 13.1 (7.06)
DLQI--Median [Median (Full Range); unit: Units on a scale] — The Dermatology Life Quality Index (DLQI) is a skin disease-specific instrument designed to assess the impact of the disease on a subject's quality of life. The scale range is 0 to 30: 0-1=no effect on subject's life; 2-5=small effect; 6-10= moderate effect; 11-20=very large effect; 21-30=extremely large effect.
  Units on a scale | 16.0 [5 to 26] | 15.0 [4 to 28] | 10.0 [0 to 27] | 12.5 [0 to 28]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Percentage of Subjects With ≥ 75% Decrease or ≥ 50% Decrease in PASI Score at EOT---ITT Population
Description: Percentage of available subjects who achieved at least a 75% reduction (PASI 75) or at least a 50% reduction from baseline in Psoriasis Area and Severity Index (PASI) score after 12 weeks of treatment with belumosudil or at the end of treatment with belumosudil in the Intent-to-Treat Population.
  [The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign is assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.]
Time Frame: 12 weeks
Population: Intent-to-Treat (ITT) Population: All subjects enrolled in study
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Groups:
- Overall (All Subjects): Belumosudil 400 mg QD + 200 mg QD + 400 mg BID for 12 weeks
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
Number analyzed (Participants) | 12 | 12 | 11 | 35
Percentage of participants (%)
  ≥ 75% Reduction from Baseline | 16.7 [2.1 to 48.4] | 8.3 [0.2 to 38.5] | 9.1 [0.2 to 41.3] | 11.4 [3.2 to 26.7]
  ≥ 50% Reduction from Baseline | 41.7 [15.2 to 72.3] | 50.0 [21.1 to 78.9] | 18.2 [2.3 to 51.8] | 37.1 [21.5 to 55.1]

2. Primary Outcome: Efficacy: Percentage of Subjects With ≥ 75% Decrease or ≥ 50% Decrease With PASI Score at EOT---Evaluable Population
Description: Percentage of available subjects who achieved at least a 75% reduction and a 50% reduction from baseline in Psoriasis Area and Severity Index score at end of treatment with belumosudil in the Evaluable Population.
  [The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign is assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.]
Time Frame: 12 weeks
Population: Evaluable Population: Subjects who receive at least 80% of the expected amount of study drug if the subject had completed the study
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
Number analyzed (Participants) | 12 | 7 | 7 | 26
Percentage of participants (%)
  ≥ 75% Reduction from Baseline | 16.7 [2.1 to 48.4] | 14.3 [0.4 to 57.9] | 14.3 [0.4 to 57.9] | 15.4 [4.4 to 34.9]
  ≥ 50% Reduction from Baseline | 41.7 [15.2 to 72.3] | 71.4 [29.0 to 96.3] | 28.6 [3.7 to 71.0] | 46.2 [26.6 to 66.6]

3. Primary Outcome: Safety: Percentage of Subjects With AEs by Severity and Relationship to Belumosudil--ITT Population
Description: Percentage of subjects who had an adverse event by severity in the Intent-to-Treat Population: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death.
  Percentage of subjects who had an adverse event by relationship to belumosudil in the Intent-to-Treat Population as assessed by the investigator: definitely related, probably related, possibly related, and not related to belumosudil.
Time Frame: 12 weeks
Population: ITT Population: All enrolled subjects
Measure: Number; unit: Percentage of participants (%)
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
Number analyzed (Participants) | 13 | 13 | 12 | 38
Percentage of participants (%)
  All AEs | 12 | 11 | 8 | 31
  Grade 1 (Mild) | 69.2 | 46.2 | 33.3 | 50.0
  Grade 2 (Moderate) | 69.2 | 46.2 | 50.0 | 55.3
  Grade 3 (Severe) | 7.7 | 7.7 | 8.3 | 7.9
  Grade 4 (Life-threatening) | 7.7 | 0 | 0 | 2.6
  Grade 5 (Death) | 0 | 0 | 0 | 0
  Related to KD025 | 38.5 | 23.1 | 58.3 | 39.5
  Grade 3, 4, or 5 Related to KD025 | 0 | 7.7 | 0 | 2.6

4. Secondary Outcome: Efficacy: Mean Change in PASI Score at 12 Weeks From Baseline--ITT Population
Description: Mean change in Psoriasis Area and Severity Index score after 12 weeks of treatment or End of Treatment with KD025 from baseline in the Intent-to-Treat Population.
  [The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign is assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.] Negative mean change is favorable; positive mean change is unfavorable
Time Frame: 12 weeks
Population: Intent-to-Treat (ITT) Population: All enrolled subjects
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
Number analyzed (Participants) | 12 | 12 | 11 | 35
Score on a scale
  End of Treatment (or 12 Weeks) | 12.4 [7.9 to 17.0] | 10.3 [7.0 to 13.6] | 14.4 [8.8 to 19.9] | 12.3 [9.9 to 14.7]
  Change from Baseline at End of Treatment | -8.8 [-16.5 to -1.1] | -6.0 [-9.5 to -2.4] | -4.8 [-8.9 to -0.7] | -6.6 [-9.5 to -3.7]
Statistical Analysis 1: Comparison: 400 mg QD; Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change in Cohort 400 mg QD PASI from baseline to Week 12; p = 0.0282, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 2: Comparison: 200 mg BID; Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change in Cohort 200 mg BID PASI from baseline to Week 12; p = 0.0035, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 3: Comparison: 400 mg BID; Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change in Cohort 400 mg BID PASI from baseline to Week 12; p = 0.0261, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 4: Comparison: Overall (All Subjects); Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change for all subjects' PASI from baseline to Week 12; p < 0.0001, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed

5. Secondary Outcome: Efficacy: Mean Change in PASI Score at 12 Weeks From Baseline--Evaluable Population
Description: Mean change in Psoriasis Area and Severity Index score after 12 weeks of treatment or end of treatment with belumosudil from baseline in the Evaluable Population.
  [The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign is assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.] Negative mean change is favorable; positive mean change is unfavorable
Time Frame: 12 weeks
Population: Intent-to-Treat (ITT) Population: All enrolled subjects
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
Number analyzed (Participants) | 12 | 7 | 7 | 26
Score on a scale
  12 Weeks | 12.4 [7.9 to 17.0] | 7.6 [5.6 to 9.6] | 15.5 [5.8 to 25.1] | 12.0 [8.9 to 15.0]
  Change from Baseline at 12 Weeks | -8.8 [-16.5 to -1.1] | -7.9 [-11.9 to -3.9] | -5.9 [-12.5 to 0.7] | -7.8 [-11.4 to -4.1]
Statistical Analysis 1: Comparison: 400 mg QD; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.0282, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 2: Comparison: 200 mg BID; Test type: Other — [test comment as in outcome 4, analysis 2]; p = 0.0029, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 3: Comparison: 400 mg BID; Test type: Other — [test comment as in outcome 4, analysis 3]; p = 0.0703, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 4: Comparison: Overall (All Subjects); Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change of all subjects' PASI from baseline to Week 12; p = 0.0002, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed

6. Secondary Outcome: Efficacy: Percentage of Subjects With a Decrease in PASI After 4 Weeks---ITT Population
Description: The percentage of subjects who exhibit any decrease in the Psoriasis Area and Severity Index score from baseline after 4 weeks of treatment with belumosudil in the Intent-to-Treat Population.
  [The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign is assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.]
Time Frame: 4 weeks
Population: Intent-to-Treat (ITT) Population: All enrolled subjects
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
Number analyzed (Participants) | 13 | 12 | 12 | 37
Percentage of participants (%) | 76.9 [46.2 to 95.0] | 66.7 [34.9 to 90.1] | 58.3 [27.7 to 84.8] | 67.6 [50.2 to 82.0]

7. Secondary Outcome: Efficacy: Percentage of Subjects With a Decrease in PASI Score After 8 Weeks---ITT Population
Description: The percentage of subjects who exhibit any decrease in the Psoriasis Area and Severity Index score from baseline after 8 weeks of treatment with belumosudil in the Intent-to-Treat Population.
  [The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign is assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.]
Time Frame: 8 weeks
Population: Intent-to-Treat (ITT) Population: All enrolled subjects
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
Number analyzed (Participants) | 12 | 9 | 7 | 28
Percentage of participants (%) | 83.3 [51.6 to 97.9] | 100 [66.4 to 100] | 85.7 [42.1 to 99.6] | 89.3 [71.8 to 97.7]

8. Secondary Outcome: Efficacy: Percentage of Subjects With a Decrease in PASI Score at EOT---ITT Population
Description: The percentage of subjects who exhibit any decrease in the Psoriasis Area and Severity Index score from baseline at the end of treatment with belumosudil in the Intent-to-Treat Population.
  [The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign is assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.]
Time Frame: 12 weeks
Population: Intent-to-Treat (ITT) Population: All enrolled subjects
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
Number analyzed (Participants) | 12 | 12 | 11 | 35
Percentage of participants (%) | 75.0 [42.8 to 94.5] | 75.0 [42.8 to 94.5] | 81.8 [48.2 to 97.7] | 77.1 [59.9 to 89.6]

9. Secondary Outcome: Efficacy: Percentage of Subjects With a Decrease in PASI Score After 4 Weeks, 8 Weeks, and 12 Weeks---Evaluable Population
Description: The percentage of subjects who exhibit any decrease in the Psoriasis Area and Severity Index score from baseline after 4 weeks, 8 weeks, and 12 weeks of treatment with belumosudil in the Evaluable Population.
  [The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign is assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.]
Time Frame: 12 weeks
Population: Evaluable Population: Subjects who received at least 80% of the expected amount study drug if the subject had completed the study
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
Number analyzed (Participants) | 12 | 7 | 7 | 26
Percentage of participants (%)
  4 Weeks | 75.0 [42.8 to 94.5] | 85.7 [42.1 to 99.6] | 71.4 [29.0 to 96.3] | 76.9 [56.4 to 91.0]
  8 Weeks | 83.3 [51.6 to 97.9] | 100 [59.0 to 100] | 85.7 [42.1 to 99.6] | 88.5 [69.8 to 97.6]
  12 Weeks | 75.0 [42.8 to 94.5] | 100 [59.0 to 100] | 85.7 [42.1 to 99.6] | 84.6 [65.1 to 95.6]

10. Secondary Outcome: Efficacy: Mean Change in PASI Score After 4 Weeks---ITT Population
Description: Mean change in the Psoriasis Area and Severity Index score from baseline after 4 weeks of treatment with belumosudil in the Intent-to-Treat Population.
  [The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign is assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.] Negative mean change is favorable; positive mean change is unfavorable
Time Frame: 4 weeks
Population: Intent-to-Treat (ITT) Population: All enrolled subjects
Measure: Number (95% Confidence Interval); unit: Score on a scale
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
Number analyzed (Participants) | 13 | 12 | 12 | 37
Score on a scale | -4.7 [-7.8 to -1.6] | -2.6 [-5.3 to 0] | -2.3 [-5.5 to 1.0] | -3.2 [-4.8 to -1.6]
Statistical Analysis 1: Comparison: 400 mg QD; Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change in Cohort 400 mg QD from baseline to Week 4; p = 0.0064, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 2: Comparison: 200 mg BID; Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change in Cohort 200 mg BID from baseline to Week 4; p = 0.0479, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 3: Comparison: 400 mg BID; Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change in Cohort 400 mg BID from baseline to Week 4; p = 0.1513, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 4: Comparison: Overall (All Subjects); Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change Overall from baseline to Week 4; p = 0.0002, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed

11. Secondary Outcome: Efficacy: Mean Change in PASI Score After 8 Weeks---ITT Population
Description: Mean change in the Psoriasis Area and Severity Index score from baseline after 8 weeks of treatment with belumosudil in the Intent-to-Treat Population.
  [The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign is assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.] Negative mean change is favorable; positive mean change is unfavorable
Time Frame: 8 weeks
Population: Intent-to-Treat (ITT) Population: All enrolled subjects
Measure: Number (95% Confidence Interval); unit: Score on a scale
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
Number analyzed (Participants) | 12 | 9 | 7 | 28
Score on a scale | -8.6 [-15.0 to -2.1] | -6.4 [-9.6 to -3.2] | -4.7 [-10.0 to 0.6] | -6.9 [-9.8 to -4.0]
Statistical Analysis 1: Comparison: 400 mg QD; Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change in Cohort 400 mg QD from baseline to Week 8; p = 0.0137, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 2: Comparison: 200 mg BID; Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change in Cohort 200 mg BID from baseline to Week 8; p = 0.0017, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 3: Comparison: 400 mg BID; Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change in Cohort 400 mg BID from baseline to Week 8; p = 0.0743, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 4: Comparison: Overall (All Subjects); Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change Overall from baseline to Week 8; p < 0.0001, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed

12. Secondary Outcome: Efficacy: Mean Change in PASI Score at 4 and 8 Weeks---Evaluable Population
Description: Mean change in the Psoriasis Area and Severity Index score from baseline after 4 and 8 weeks of treatment with belumosudil in the Evaluable Population.
  [The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign is assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.] Negative mean change is favorable; positive mean change is unfavorable
Time Frame: 8 weeks
Population: Evaluable Population: Subjects who received at least 80% of the expected amount of study drug if the subject had completed the study
Measure: Number (95% Confidence Interval); unit: Score on a scale
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
Number analyzed (Participants) | 12 | 7 | 7 | 26
Score on a scale
  4 Weeks | -4.4 [-7.8 to -1.1] | -3.5 [-7.2 to 0.2] | -2.7 [-8.1 to 2.7] | -3.7 [-5.7 to -1.7]
  8 Weeks | -8.6 [-15.0 to -2.1] | -6.8 [-10.9 to -2.7] | -4.7 [-10.0 to 0.6] | -7.1 [-10.2 to -3.9]
Statistical Analysis 1: Comparison: 400 mg QD; Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change in Cohort 400 mg QD from baseline to 4 weeks; p = 0.0140, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 2: Comparison: 200 mg BID; Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change in Cohort 200 mg BID from baseline to 4 weeks; p = 0.0620, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 3: Comparison: 400 mg BID; Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change in 400 mg BID from baseline to 4 weeks; p = 0.2620, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 4: Comparison: Overall (All Subjects); Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change of all subjects from baseline to 4 weeks; p = 0.0008, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 5: Comparison: 400 mg QD; Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change in Cohort 400 mg QD from baseline to 8 weeks; p = 0.0137, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 6: Comparison: 200 mg BID; Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change in Cohort 200 mg BID from baseline to 8 weeks; p = 0.0064, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 7: Comparison: 400 mg BID; Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change in Cohort 400 mg BID from baseline to 8 weeks; p = 0.0743, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 8: Comparison: Overall (All Subjects); Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change of all subjects from baseline to 8 weeks; p < 0.0001, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed

13. Secondary Outcome: Efficacy: Percentage of Subjects With Improvement in PGA af 4 Weeks---ITT Population
Description: Percentage of subjects evaluated by the Physician Global Assessment who improve (excellent, good, or fair) from baseline after 4 weeks of treatment with belumosudil in the Intent-to-Treat Population.
  The relative PGA documents the physician's assessment of the subject's psoriasis status. Consideration was given to the percent of body involvement as well as overall induration, scaling, and erythema. The PGA was assessed relative to baseline condition and was defined as: (1) clear; (2) excellent; (3) good; (4) fair; (5) poor; and (6) worse PGA improvement is defined as the categorical change from baseline: Clear = 100% improvement; Excellent = 75% to 99% improvement; Good = 50% to 74% improvement; Fair = 25% to 49% improvement
Time Frame: 4 weeks
Population: Intent-to-Treat (ITT) Population: All enrolled subjects
Measure: Number; unit: Percentage of participants
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
Number analyzed (Participants) | 13 | 12 | 12 | 37
Percentage of participants
  Clear/Excellent (75% to 100% Improvement) | 0 | 0 | 0 | 0
  Good (50% to 74% Improvement) | 7.7 | 8.3 | 8.3 | 8.1
  Fair (25% to 49% Improvement) | 46.2 | 58.3 | 41.7 | 48.6

14. Secondary Outcome: Efficacy: Percentage of Subjects With Improvement in PGA af 8 Weeks---ITT Population
Description: Percentage of subjects evaluated by the Physician Global Assessment who improve (excellent, good, or fair) from baseline after 8 weeks of treatment with belumosudil in the Intent-to-Treat Population.
  The relative PGA documents the physician's assessment of the subject's psoriasis status. Consideration was given to the percent of body involvement as well as overall induration, scaling, and erythema. The PGA was assessed relative to baseline condition and was defined as: (1) clear; (2) excellent; (3) good; (4) fair; (5) poor; and (6) worse.
  PGA improvement is defined as the categorical change from baseline: Clear = 100% improvement; Excellent = 75% to 99% improvement; Good = 50% to 74% improvement; Fair = 25% to 49% improvement
Time Frame: 8 weeks
Population: Intent-to-Treat (ITT) Population: All enrolled subjects
Measure: Number; unit: Percentage of participants
Groups:
- 400 mg QD: Belumosudl 400 mg PO QD for 12 weeks
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
Number analyzed (Participants) | 12 | 9 | 7 | 28
Percentage of participants
  Clear/Excellent (75% to 100% Improvement) | 8.3 | 0 | 0 | 3.6
  Good (50% to 74% Improvement) | 25.0 | 11.1 | 14.3 | 17.9
  Fair (25% to 49% Improvement) | 25.0 | 88.9 | 42.9 | 50.0

15. Secondary Outcome: Efficacy: Percentage of Subjects With Improvement in PGA af EOT--ITT Population
Description: Percentage of subjects evaluated by the Physician Global Assessment who improve (excellent, good, or fair) from baseline after 12 weeks of treatment with belumosudil or at the end of treatment (EOT) in the Intent-to-Treat Population.
  The relative PGA documents the physician's assessment of the subject's psoriasis status. Consideration was given to the percent of body involvement as well as overall induration, scaling, and erythema. The PGA was assessed relative to baseline condition and was defined as: (1) clear; (2) excellent; (3) good; (4) fair; (5) poor; and (6) worse.
  PGA improvement is defined as the categorical change from baseline: Clear = 100% improvement; Excellent = 75% to 99% improvement; Good = 50% to 74% improvement; Fair = 25% to 49% improvement
Time Frame: 12 weeks
Population: Intent-to-Treat (ITT) Population: All enrolled subjects
Measure: Number; unit: Percentage of participants
Groups:
- Overall (All Subjects): Belumosudil 400 mg PO QD + 200 mg PO QD + 400 mg PO BID for 12 weeks
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
Number analyzed (Participants) | 12 | 12 | 11 | 35
Percentage of participants
  Clear/Excellent (75% to 100% Improvement) | 0 | 0 | 0 | 0
  Good (50% to 74% Improvement) | 33.3 | 25.0 | 18.2 | 25.7
  Fair (25% to 49% Improvement) | 33.3 | 50.0 | 36.4 | 40.0

16. Secondary Outcome: Efficacy: Percentage of Subjects With Improvement in PGA af 4, 8, and 12 Weeks---Evaluable Population
Description: Percentage of subjects evaluated by the Physician Global Assessment who improve (excellent, good, or fair) from baseline after 4 weeks, after 8 weeks, and after 12 week of treatment with belumosudil in the Evaluable Population.
  The relative PGA documents the physician's assessment of the subject's psoriasis status. Consideration was given to the percent of body involvement as well as overall induration, scaling, and erythema. The PGA was assessed relative to baseline condition and was defined as: (1) clear; (2) excellent; (3) good; (4) fair; (5) poor; and (6) worse.
  PGA improvement is defined as the categorical change from baseline: Clear = 100% improvement; Excellent = 75% to 99% improvement; Good = 50% to 74% improvement; Fair = 25% to 49% improvement.
Time Frame: 12 weeks
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
Number analyzed (Participants) | 12 | 7 | 7 | 26
Percentage of participants
  4 Weeks: Clear/Excellent | 0 | 0 | 0 | 0
  4 Weeks: Good | 8.3 | 0 | 14.3 | 7.7
  4 Weeks: Fair | 41.7 | 85.7 | 42.9 | 53.8
  8 Weeks: Clear/Excellent | 8.3 | 0 | 0 | 3.8
  8 Weeks: Good | 25.0 | 0 | 14.3 | 15.4
  8 Weeks: Fair | 25.0 | 100 | 42.9 | 50.0
  12 Weeks: Clear/Excellent | 0 | 0 | 0 | 0
  12 Weeks: Good | 33.3 | 14.3 | 28.6 | 26.9
  12 Weeks: Fair | 33.3 | 85.7 | 28.6 | 46.2

17. Secondary Outcome: Efficacy: Mean Changes in DLQI at EOT--ITT Population
Description: Mean changes in the Dermatology Life Quality Index from baseline after 12 weeks of treatment with belumosudil or end of treatment with KD025 in the Intent-to-Treat Population [The Dermatology Life Quality Index (DLQI) is a skin disease-specific instrument designed to assess the impact of the disease on a subject's quality of life. The scale range is 0 to 30: 0-1=no effect on subject's quality of life; 2-5=small effect; 6-10= moderate effect; 11-20=very large effect; 21-30=extremely large effect.] Negative mean change is favorable; positive mean change is unfavorable
Time Frame: 12 weeks
Population: Intent-to-Treat: All enrolled subjects.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
Number analyzed (Participants) | 12 | 12 | 11 | 35
Score on a scale | -4.9 (4.68) | -5.1 (5.35) | -2.5 (4.50) | -4.2 (4.86)
Statistical Analysis 1: Comparison: 400 mg QD; Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change in Cohort 400 mg QD from baseline to 12 weeks; p = 0.004, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 2: Comparison: 200 mg BID; Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change in Cohort 200 mg BID from baseline to 12 weeks; p = 0.007, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 3: Comparison: 400 mg BID; Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change in Cohort 400 mg BID from baseline to 12 weeks; p = 0.090, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 4: Comparison: Overall (All Subjects); Test type: Other — No control group was used. Paired t-testing was used to determine the statistical significance of the mean change Overall from baseline to 12 weeks; p < 0.001, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed

18. Secondary Outcome: Efficacy: Mean Changes in DLQI at 12 Weeks--Evaluable Population
Description: Mean changes in the Dermatology Life Quality Index (DLQI) score from baseline after 12 weeks of treatment with belumosudil in the Evaluable Population.
  [The Dermatology Life Quality Index (DLQI) is a skin disease-specific instrument designed to assess the impact of the disease on a subject's quality of life. The scale range is 0 to 30: 0-1=no effect on subject's quality of life; 2-5=small effect; 6-10= moderate effect; 11-20=very large effect; 21-30=extremely large effect.] Negative mean change is favorable; positive mean change is unfavorable.
Time Frame: 12 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
Number analyzed (Participants) | 12 | 7 | 7 | 26
Score on a scale | -4.9 (4.68) | -6.3 (5.82) | -2.3 (2.93) | -4.6 (4.71)
Statistical Analysis 1: Comparison: 400 mg QD; Test type: Superiority; p = 0.004, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 2: Comparison: 200 mg BID; Test type: Superiority; p = 0.029, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 3: Comparison: 400 mg BID; Test type: Superiority; p = 0.084, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed
Statistical Analysis 4: Comparison: Overall (All Subjects); Test type: Superiority; p < 0.001, t-test, 2 sided — Statistical significance was set at p ≤ 0.05. No adjustments for multiplicity were made. Missing data were not imputed

19. Secondary Outcome: Pharmacokinetics: Cmax of Parent Drug KD025, KD025m1, and KD025m2
Description: Maximum concentration (Cmax) of Parent drug (KD0250), Metabolite 1 (KD025m1), and Metabolite 2 (KD025m2)
Time Frame: 24 hours
Population: PK Population: Subjects received at least 1 dose of study drug and had at least 1 post-dose PK sample drawn.
  Note: Not all subjects had all data available for PK parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 400 mg QD: Belumosudil 400 mg administered QD (once daily)
- 200 mg BID: Belumosudil 200 mg administered PO BID (twice daily)
Arm/Group | 400 mg QD | 200 mg BID
Number analyzed (Participants) | 7 | 6
ng/mL
  KD025 | 3140 (1760) | 1770 (1190)
  KD025m1: number analyzed (Participants) | 6 | 4
  KD025m1 | 23.2 (9.66) | 22.8 (15.3)
  KD025m2: number analyzed (Participants) | 6 | 6
  KD025m2 | 632 (278) | 203 (204)

20. Secondary Outcome: Pharmacokinetics: AUC of Parent Drug KD025, KD025m1, and KD025m2
Description: Area Under Concentration Time Curve (AUC) for Parent Drug KD025, Metabolite 1 (KD025m1), and Metabolite 2 (KD025m2):
  AUC(0-12) = AUC from predose to 12 hours post-dose AUC(0-24) = AUC from predose to 24 hours post-dose AUC(0-t) = AUC from predose to a given time "t" post-dose
Time Frame: 24 hours
Population: PK Population: Subjects received at least 1 dose of study drug and had at least 1 post-dose PK sample drawn.
  Note: KD025m2 did not have AUC(0-12) or AUC(0-24) available. Not all subjects had all PK measurements. AUC(0-12) and AUC(0-24) for KD025m1 were not calculable.
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | 400 mg QD | 200 mg BID
Number analyzed (Participants) | 7 | 6
hour*ng/mL
  KD025: AUC(0-12) | 16200 (8910) | 9150 (5950)
  KD025m2: AUC(0-12): number analyzed (Participants) | 6 | 6
  KD025m2: AUC(0-12) | 2300 (907) | 757 (823)
  KD025: AUC(0-24) | 18800 (10600) | 21800 (13900)
  KD025m2: AUC(0-24): number analyzed (Participants) | 5 | 6
  KD025m2: AUC(0-24) | 2510 (1180) | 1790 (1850)
  KD025: AUC(0-t) | 18800 (10600) | 25100 (14800)
  KD025m1: AUC(0-t): number analyzed (Participants) | 3 | 1
  KD025m1: AUC(0-t) | 93.4 (18.1) | 250 (0)
  KD025m2: AUC(0-t): number analyzed (Participants) | 6 | 6
  KD025m2: AUC(0-t) | 2550 (1080) | 1960 (1950)

21. Secondary Outcome: Pharmacokinetics: t(1/2) of KD025
Description: Half-life (t[1/2]) of Parent drug (KD025)
Time Frame: 24 hours
Population: Subjects received at least 1 dose of study drug and had at least 1 post-dose PK sample drawn.
  One subject in 200 mg BID cohort did not have t(1/2) data available.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | 400 mg QD | 200 mg BID
Number analyzed (Participants) | 7 | 5
Hours | 8.00 (2.47) | 5.13 (1.12)

22. Secondary Outcome: Pharmacokinetics: MR C(Max) and MR AUC(0-t) for KD025m1 and KD025m2
Description: Metabolite-to-parent ratio of maximum concentration (MR C[max]) and metabolite-to-parent ratio of the area under concentration time curve from pre-dose to a given time "t" for Metabolite 1 (KD025m1) and Metabolite 2 (KD025m2)
Time Frame: 24 hours
Population: The metabolite-to-parent ratio is not applicable to parent drug KD025. Not all subjects had data for all PK parameters.
Measure: Mean (Standard Deviation); unit: Number (ratio)
Arm/Group | 400 mg QD | 200 mg BID
Number analyzed (Participants) | 7 | 6
Number (ratio)
  KD025m1: MR C(max): number analyzed (Participants) | 6 | 4
  KD025m1: MR C(max) | 0.00736 (0.00272) | 0.00984 (0.00287)
  KD025m2: MR C(max): number analyzed (Participants) | 6 | 6
  KD025m2: MR C(max) | 0.199 (0.0794) | 0.101 (0.0469)
  KD025m1: MR AUC(0-t): number analyzed (Participants) | 3 | 1
  KD025m1: MR AUC(0-t) | 0.00458 (0.00253) | 0.00577 (0)
  KD025m2: MR AUC(0-t): number analyzed (Participants) | 6 | 6
  KD025m2: MR AUC(0-t) | 0.133 (0.0449) | 0.0719 (0.0336)

ADVERSE EVENTS:
Time Frame: Screening Period ≤ 4 week Screening Period + 12-week Treatment Period + 30-day Follow-up = Up to 20 weeks
Arm/Group | 400 mg QD | 200 mg BID | 400 mg BID | Overall (All Subjects)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/12 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/12 | 0/38
Other Adverse Events (participants affected / at risk) | 12/13 | 11/13 | 8/12 | 31/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 400 mg QD (N=13) | 200 mg BID (N=13) | 400 mg BID (N=12) | Overall (All Subjects) (N=38)
Liver function test abnormal (Investigations) | 1 (1) | 1 (3) | 1 (2) | 3 (6)
Transaminases increased (Investigations) | 1 (5) | 1 (1) | 0 (0) | 2 (6)
Alanine aminotransaminase (ALT) increased (Investigations) | 1 (1) | 0 (0) | 4 (4) | 5 (5)
Aspartate aminotransferase (AST) increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Oral herpes (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tonsilitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Paransal sinus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Edema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anorgasmia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding results. The sponsor cannot require changes to the study results in the communication except to remove sponsor's confidential information. Sponsor cannot unilaterally extend the embargo.